CLINICAL TRIAL: NCT04119453
Title: A Phase 2 Open-Label, Multicenter, Study to Evaluate the Efficacy and Safety of Rivoceranib in Subjects With Recurrent or Metastatic Adenoid Cystic Carcinoma of All Anatomic Sites of Origin
Brief Title: A Study to Evaluate the Efficacy and Safety of Rivoceranib in Participants With Recurrent or Metastatic Adenoid Cystic Carcinoma (ACC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The RM-202 study was terminated by the Sponsor due to redirection of the rivoceranib development plan.
Sponsor: Elevar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RM-202
Record Dates: First submitted 2019-09-24; First posted 2019-10-08 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Adenoid Cystic Carcinoma
MeSH Terms: conditions — Carcinoma, Adenoid Cystic | interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rivoceranib (Experimental): Participants will receive an oral dose of rivoceranib once per day during 28-day cycles.
  Interventions: Drug: Rivoceranib

INTERVENTIONS:
Drug: Rivoceranib — Film-coated tablets
  Other Names: Apatinib, Apatinib Mesylate

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of rivoceranib in adult participants with recurrent or metastatic ACC. All participants may remain on treatment until occurrence of disease progression, unacceptable toxicity, death, the withdrawal of consent from treatment, lost to follow-up or study termination by the Sponsor. When a participant discontinues rivoceranib for any reason, the participant will enter the 24 month survival follow up period until withdrawal of consent from the study, lost to follow up, end of the study or death, whichever occurs earlier.

The maximum duration of the study is estimated to be 48 months and includes screening, treatment, and follow-up phases.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed metastatic/recurrent ACC not amenable to potentially curative surgery or radiotherapy
2. Evidence of disease progression by RECIST v1.1

   Note: Disease progression is defined as one of the following occurring within the 6 months prior to study entry:
   1. At least a 20% increase in radiologically or clinically measurable lesions
   2. Appearance of any new lesions
3. Presence of at least one measurable target lesion which is evaluable by RECIST v1.1 criteria
4. Participants are eligible if central nervous system (CNS) metastases have been treated and participants are neurologically returned to baseline or neurologically stable in the opinion of Investigator (except for residual signs or symptoms related to the CNS treatment) for at least 4 weeks prior to first dose of study drug administration. In addition, participants must be either off corticosteroids, or on a stable dose or decreasing dose of <20 milligrams (mg) daily prednisone or prednisone equivalent.

   Note: Only participants with a known history or indication of CNS disease are required to have CNS imaging prior to study entry
5. Adequate organ and marrow function within 14 days prior to the first dose of rivoceranib administration, defined as:

   1. Absolute neutrophil count ≥1500/microliters (μL)
   2. Platelet count ≥100,000/μL
   3. Serum bilirubin ≤1.5× upper limit of normal (ULN)
   4. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3.0×ULN (≤5.0×ULN, if with liver metastasis)
   5. Estimated Creatinine Clearance >50 milliliters (mL)/minute (min) (Cockcroft-Gault)
   6. Partial thromboplastin time (PTT), prothrombin time (PT) and international normalized ratio (INR) ≤1.5×ULN
   7. Hemoglobin ≥9.0 grams (g)/deciliter (dL)
6. Urinary protein <2+ on dipstick or routine urinalysis. If urine dipstick or routine analysis indicates proteinuria ≥2+, a 24-hour urine or urine protein/creatinine ratio must be collected and must demonstrate <2 g of protein in 24 hours.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
8. The ability to understand and the willingness to sign a written informed consent
9. Female participants who are of non-reproductive potential (that is, post-menopausal by history - no menses for ≥1 year; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy). Female participants of childbearing potential must have a negative serum pregnancy test within 72 hours prior to the first dose of rivoceranib.
10. Male and female participants of reproductive potential who agree to use both a highly effective method of birth control (for example, implants, injectables, combined oral contraceptives, some intrauterine devices, complete abstinence, or sterilized partner) and a barrier method (for example condoms, cervical ring, sponge, etc.) during the period of therapy and for 30 days after the final dose of rivoceranib. Female participants should also refrain from breastfeeding and egg donation and males should refrain from sperm donation throughout this period
11. QTc interval <480 milliseconds (ms) (Common Terminology Criteria for Adverse Events [CTCAE] Grade 1) using Fredericia's QT correction formula

Exclusion Criteria:

1. Previous treatment with rivoceranib
2. Known hypersensitivity to rivoceranib or components of the formulation
3. Packed red blood cell transfusion or erythropoietin therapy within 14 days prior to the first dose of rivoceranib administration
4. History of another malignancy within 3 years prior to enrollment. A participant with the following malignancies is eligible for this study if, surgically and medically treated and in the opinion of the investigator, they do not pose a significant risk to life expectancy or not likely to recur within 3 years:

   1. Carcinoma of the skin without melanomatous features
   2. Curatively treated cervical carcinoma in situ
   3. Bladder tumors considered superficial such as noninvasive (T1a) and carcinoma in situ (Tis)
   4. Thyroid papillary cancer with prior treatment
   5. Prostate cancer which has been surgically or medically treated
5. Prior chemotherapy, radiation therapy or major surgery within 4 weeks prior to rivoceranib administration or presence of any nonhealing wound (procedures such as catheter placement are not considered to be major surgery). Prior immunotherapy within 12 weeks prior to first dose of study drug. Palliative radiotherapy to non-target lesions within 2 weeks prior to rivoceranib administration or biopsy any time prior to rivoceranib administration is permitted.
6. Prior tyrosine kinase inhibitor therapy targeting vascular endothelial growth factor receptors (VEGFR), within 5 half-lives prior to rivoceranib administration
7. Participants who have not recovered to ≤Grade 1 from prior tyrosine kinase inhibitor-related adverse events
8. History of uncontrolled hypertension based on Investigator's clinical judgement (consistent blood pressure readings ≥140/90 millimeters of mercury [mmHg] and/or change in antihypertensive medication within 7 days prior to rivoceranib administration)
9. History of severe adverse events including uncontrolled hypertension or other common anti-angiogenesis class drug effects (for example, ramucirumab) that may indicate a higher risk to the safety of the participant if provided further anti-angiogenesis treatment, in the investigator's opinion.
10. History of vascular disease including arterial or venous embolic events (pulmonary embolism), other than hypertension, within the last 3 months prior to treatment with rivoceranib (for example, hypertensive crisis, hypertensive encephalopathy, stroke or transient ischemic attack [TIA], or significant peripheral vascular diseases) that, in the investigator's opinion, may pose a risk to the participant on vascular endothelial growth factor (VEGF) inhibitor therapy.
11. History of bleeding diathesis or clinically significant bleeding within 14 days prior to treatment with rivoceranib
12. History of clinically significant thrombosis within 3 months prior to treatment with rivoceranib that, in the investigator's opinion, may place the participant at risk of side effects from anti-angiogenesis products
13. Therapy with systemic anticoagulant or antithrombotic agents within 7 days prior to treatment with rivoceranib that in the investigator's opinion could interfere with clotting. The maximum allowable daily dose of aspirin is 325 mg.
14. Gastrointestinal malabsorption, or any other condition that in the opinion of the investigator might affect the absorption of rivoceranib
15. History of clinically significant glomerulonephritis, biopsy-proven tubulointerstitial nephritis, crystal nephropathy, or other renal insufficiencies
16. An uncontrolled intercurrent illness including, but not limited to any of the following:

    1. Ongoing or active infection (including minor localized infections) requiring oral or intravenous treatment
    2. Symptomatic class 3 or 4 congestive heart failure, defined as a clinical syndrome resulting from any structural or functional cardiac disorder that impairs the ability of the ventricle to fill with or eject blood
    3. Unstable angina pectoris
    4. Cardiac arrhythmia
    5. Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the participant's safety or study endpoints
17. A female participant who is pregnant or breast-feeding
18. Psychiatric illness/social situations that would limit compliance with study requirements
19. History of drug or alcohol abuse within the past 5 years
20. Known seropositive requiring anti-viral therapy for human immunodeficiency virus (HIV) infection
21. Known seropositive requiring antiviral therapy for hepatitis B virus (HBV) infection OR evidence of active hepatitis B infection by detectable viral load if the antibody tests are positive NOTE: A positive hepatitis B core antibody (HBcAb) participant with an undetectable surface antigen and negative hepatitis B deoxyribonucleic acid (DNA) test (for example, polymerase chain reaction [PCR] test) can be enrolled.
22. Known seropositive requiring antiviral therapy for hepatitis C virus (HCV) infection OR participants with positive hepatitis C virus antibody NOTE: A positive Anti-HCV participant with an undetectable/negative hepatitis C ribonucleic acid (RNA) test can be enrolled.
23. Participation in another clinical study with any investigational medication or product administered within ≤28 days prior to first dose of rivoceranib
24. Participants unable or unwilling to discontinue excluded medications for at least 5 half-lives prior to first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR): Percentage of Participants who Achieve Confirmed Complete Response (CR) or Partial Response (PR) | Up to 48 months
  ORR per the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 by investigator/institutional assessment.
Objective Response Rate (ORR): Percentage of Participants who Achieve Confirmed Complete Response (CR) or Partial Response (PR) | Up to 48 months
  ORR per the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 by Independent Central Review.

SECONDARY OUTCOMES:
Overall Survival (OS) at 1 Year and 2 Years | Years 1 and 2
Duration of Response (DoR) | Up to 48 months
  DoR per RECIST 1.1 by investigator/institutional assessment.
Duration of Response (DoR) | Up to 48 months
  DoR per RECIST 1.1 by Independent Central Review.
Progression free survival (PFS) at 6 Months, 12 Months, and 2 Years | Months 6 and 12, and Year 2
  PFS per RECIST 1.1 by investigator/institutional assessment.
Progression free survival (PFS) at 6 Months, 12 Months, and 2 Years | Months 6 and 12, and Year 2
  PFS per RECIST 1.1 by Independent Central Review.
Time to progression (TTP) | Up to 48 months
  TTP per RECIST 1.1 by investigator/institutional assessment.
Time to progression (TTP) | Up to 48 months
  TTP per RECIST 1.1 by Independent Central Review.
Number of Participants With Adverse Events (AEs) | Up to 48 months

CONTACTS AND LOCATIONS:
Locations (11):
- United States (7):
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - UCSF, San Francisco, California
  - University of Colorado Denver, Denver, Colorado
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Dana-Farber Cancer Institute - Head and Neck Oncology, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
- South Korea (4):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Asan Medical Center, Seoul, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Gyeonggi-do
  - Samsung Medical Center, Seoul